CLINICAL TRIAL: NCT01044303
Title: An Exploratory, Open-Label, Single Center Study to Assess the Efficacy and Dose Titration of Enteric-Coated Mycophenolate Sodium (EC-MPS) in Reducing Donor Specific Antibody (DSA) Strength in Maintenance Kidney Transplant Recipients
Brief Title: Reducing Donor Specific Antibody (DSA) Strength in Maintenance Kidney Transplant Recipients (DSA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Paul Bolin, Chair of Internal Medicine, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A-US78T
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Transplant; Failure, Kidney
Keywords: Kidney Transplantation; Mycophenolic Acid; Donor-Specific Antibodies; Kidney Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myfortic Escalation (Experimental): Participants EC-MPS dose was escalated to a minimum daily dose of 1440mg or equivalent, with the maximum dose never exceeding the manufacturer's recommendations.
  Interventions: Drug: Myfortic Escalation

INTERVENTIONS:
Drug: Myfortic Escalation — Dose increases of 180 mg every 3 months until DSA titer is zero or until maximum tolerable dose of EC-MPS is achieved. Maximum dose will not exceed 2160 mg daily.
  Other Names: Enteric-coated mycophenolate sodium

SUMMARY:
The purpose of this study is to demonstrate that increased dosages of mycophenolic acid in maintenance kidney transplant recipients may cause a reduction in donor-specific antibodies.

DETAILED DESCRIPTION:
The development of DSA post-transplant has been associated with chronic rejection and graft failure. EC-MPS is thought to be the key drug preventing both cellular and antibody mediated rejections. Several studies have shown that recipients receiving an optimal dose of EC-MPS have fewer antibody mediated rejections and may require a lower dose of calcineurin inhibitors and/or corticosteroids thus reducing side effects and extending graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of cadaveric, living related or living unrelated kidney transplant with positive DSA titer.
* Males and females, 18-75 years of age.
* Patients currently receiving MPA (500mg to 2500 mg of CellCept daily or 360 mg to 1800 mg of myfortic daily), cyclosporine or tacrolimus with or without corticosteroids as part of their immunosuppressive regimen for at least 6 months.
* Females of childbearing potential must have a negative pregnancy test prior to enrollment. The test should be performed at baseline visit. Effective contraception must be used during the trial, and for 4 weeks following discontinuation of the study medication.
* Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion criteria:

* Multi-solid or cellular organ transplants (e.g. combined with pancreas, liver, islet, bone marrow), either concurrent or previous (with exception that a second kidney transplant is allowed).
* Evidence of graft rejection or treatment of acute rejection within 14 days prior to Baseline visit.
* Patients who have received any investigational drug within 4 weeks prior to study entry.
* Patients with thrombocytopenia (<75,000/mm3), with an absolute neutrophil count of <1,500/mm3 and/or leukocytopenia (<4,000/mm3), and/or hemoglobin <9.0 g/dL prior to enrollment.
* The presence of a severe GI disorder (such as Irritable Bowel Syndrome, Inflammatory Bowel Disease and known Peptic Ulcer Disease).
* Presence of clinically significant infection requiring continued therapy, chronic infection (e.g. HIV, Hep B and Hep C), malignancy (within last 5 years, except excised squamous or basal cell carcinoma of the skin), lymphoma or renal toxicity that would interfere with the appropriate conduct of the study.
* Evidence of severe liver disease (incl. abnormal liver profile i.e. AST, ALT or total bilirubin ≥ 3 times ULN) or severe diarrhea or active peptic ulcer disease that would interfere with the appropriate conduct of the study.
* Abnormal physical or laboratory findings of clinical significance within 2 weeks of inclusion which would interfere with the objectives of the study.
* Patients with symptoms of significant somatic or mental illness or evidence of drug and/or alcohol abuse.
* Patients receiving > 10 mg/day prednisone dose.
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures to MPA.
* Patients not making DSA antibodies.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (local); females of childbearing potential who are unwilling to use effective means of contraception and who are planning to become pregnant.
* Any other medical condition that, in the opinion of the site investigator based on recall or chart review would interfere with completing the study, including but not limited to visual problems or cognitive impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bolin, MD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolic Acid Escalation: Participants MPA dose was escalated to a minimum daily dose of 1440mg or equivalent, with the maximum dose never exceeding the manufacturer's recommendations.
  Enteric-coated mycophenolate sodium: Dose increases of 180 mg every 3 months until DSA titer is zero or until maximum tolerable dose of mycophenolic acid is achieved. Maximum dose will not exceed 2160 mg daily.
Period: Overall Study
Arm/Group | Mycophenolic Acid Escalation
Started | 32
Completed | 30
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mycophenolic Acid Escalation
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Mean Fluorescence Index (MFI) of Donor Specific Antibodies (DSA) With Increasing Doses of Enteric-Coated Mycophenolate Sodium (EC-MPS)
Time Frame: 24 months
Population: This was a pilot study to examine the effect of MPA escalation on DSA reduction.
Measure: Mean (Standard Deviation); unit: percent of MFI change
Groups:
- Mycophenolic Acid (MPA) Escalation: Patients receiving MPA (500mg to 2500mg of CellCept daily or 360mg to 1800mg myfortic daily), cyclosporine or tacrolimus with or without corticosteroids as part of their immunosuppressive regimen for at least 6 months
Arm/Group | Mycophenolic Acid (MPA) Escalation
Number analyzed (Participants) | 30
percent of MFI change | 43.1 (31.45)

2. Secondary Outcome: To Assess the Rate of Rejection, Infection and Renal Function as Mycophenolic Acid Dose is Increased.
Time Frame: 24 months
Measure: Number; unit: participants
Groups:
- Rate of Infection: Number of patients who had an infection during the course of the study.
- Rate of Rejection: Number of patients who had a rejection during the course of the study.
- Renal Function: Number of patients who had stable renal function throughout the study.
Arm/Group | Rate of Infection | Rate of Rejection | Renal Function
Number analyzed (Participants) | 30 | 30 | 30
participants | 2 | 2 | 29

ADVERSE EVENTS:
Groups:
- Adverse Events: Adverse events reported by participants during the course of the study.
Arm/Group | Adverse Events
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=30)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — One subject was hospitalized for pneumonia during the study period.
Diarrhea (Gastrointestinal disorders) | 2 (2) — There were two subjects hospitalized for Gastrointestinal complaints and diarrhea.
Pancreatitis (Endocrine disorders) | 1 (1) — One subject hospitalized for pancreatitis during the study
Sepsis (Blood and lymphatic system disorders) | 1 (1) — One subject was hospitalized for Sepsis during the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=30)
Diarrhea (Gastrointestinal disorders) | 3 (3)
CMV (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Lost to follow-up was a limitation in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No